Official Title: Text-Message-Based Depression Prevention for High-Risk Youth in the ED (iDOVE)

NCT Number: 02332239 Date of Document: 10/19/2015

# RESEARCH PLAN SPECIFIC AIMS:

A history of violence strongly correlates with adolescent depression.[1-5] Approximately 50% of teens with a history of physical peer (non-partner) violence, as compared to 5-10% of teens in the community, report depressive symptoms;[3, 6-9] and teens at with a history of peer violence are at increased risk of subsequent major depression.[10-12] Conversely, adolescents with depressive symptoms have higher rates of future peer victimization and aggression than non-depressed peers.[13-17] Peer violence and depression have mutual, reinforcing negative impacts on emotional and behavioral regulation strategies.[13, 18-20] Teens with a history of peer victimization or aggression are also at higher risk for other negative consequences, including anxiety, post-traumatic stress disorder (PTSD), risky sexual behaviors, and substance/alcohol abuse.[3, 4, 9, 21-24]

The emergency department (ED) is an ideal location to initiate interventions for high-risk adolescents. [25-27] Multi-session cognitive behavioral therapy (CBT) for teens' co-occurring depression and violence may effectively reduce depressive symptoms. [28, 29] However, many teens lack access to these services. [30] The ED is the primary source of care for most high-risk teens. [31, 32] An ED visit therefore provides an important opportunity to initiate preventive interventions, to complement existing mental health treatment or to stand alone for those who never seek formal care. [33-36] Innovative techniques are needed to engage ED patients. Most teens use text-messaging. [37] Personalized text-message interventions for adolescents, including for depression prevention, are accessible, feasible, and may be effective. [38-41]

In this K23 research plan, we will create an indicated depression prevention intervention for teens seen in the ED with depressive symptoms and a history of peer violence. Drawing on effective CBT and motivational interviewing (MI) depression and violence prevention interventions,[42-45] a brief in-person session ("ED") will introduce basic cognitive and behavioral strategies. Following ED discharge, eight weeks of tailored CBT-informed daily text messages ("text") will be sent, to enhance skills and remind participants of self-determined goals. The "ED+text" intervention may be more accessible and disseminable for this high-risk population.[46]

My long-term goal is to become an expert in easily-disseminated, technology-assisted mental health interventions for high-risk ED patients. Although such interventions may have a modest effect, I am purposely designing them to have a broad reach for the large group of ED patients who do not access any mental health care. My short-term goals, for this K23 award, are to gain training in development and analysis of technology-assisted ED depression prevention interventions, and to test the hypothesis that an "ED+text" indicated depression prevention intervention is acceptable and feasible. This study will lead to an R01 application to conduct formal efficacy testing.

We are currently completing our recruitment for, and analysis of, Aim1 (qualitative interviews to develop the intervention). THIS APPLICATION IS FOR APPROVAL OF AIMS 2 and 3.

<u>Aim 2: Refine intervention content.</u> Eligible participants will be iteratively enrolled, 4 at a time, in the "ED+text" intervention (n=16-20). Through semi-structured interviews and measures of protocol adherence, we will refine content and improve feasibility, acceptability, usability, and clarity of the intervention components.

# Aim 3: Conduct a randomized pilot trial (n=120) of the "ED+text" preventive intervention vs. enhanced usual care (attention-matched nutritional text messages).

**3a:** Primary outcomes will be intervention <u>acceptability</u> (defined as 65% enrollment rates and 80% agree/strongly agree ratings[42, 47] on the Client Satisfaction Questionnaire-8[48] and exit interviews), <u>feasibility</u> (defined as 80% completion of in-person and text-message sessions[42, 47]) and <u>fidelity</u> of in-person sessions (defined as 80% adherence to session manual[49-51]).

**3b**: *Preliminary hypothesis testing*: Although not powered to detect efficacy, we will look for a trend toward a <u>primary outcome</u> (a decrease in depressive symptoms at 8 and 16 weeks), and an exploratory <u>secondary</u> outcome (decreased number of peer fights) relative to enhanced usual care.

This proposal is <u>innovative</u>: it will develop a feasible, acceptable depression prevention intervention for a high-risk population of adolescent ED patients with a history of peer violence. It also has high <u>significance and impact</u>: utilizing the ED location, it addresses a current lack of easily-accessible preventive services and reflects NIMH Strategic Objectives 3 and 4. It will potentially lead to an efficient means to reduce depressed mood in high-risk teens with little access to traditional mental health care. If effective, this intervention will be

| translated to other at-risk patients seen in the ED. Finally, it is <u>essential for my career development</u> as an ED-based mental health intervention researcher. |
|---|

#### RESEARCH STRATEGY

(a) <u>SIGNIFICANCE</u>: Prevention of adolescent mental health disorders and peer violence are critical research goals according to Healthy People 2020, NIMH, and the Institute of Medicine. [52-55] Mood disorders are epidemic among teens, [6-8, 56] and strongly correlate with a history of physical peer violence (assault or victimization). [5, 14, 15, 57-59] Rates of youth violence are also high, [60, 61] many causing severe injury: over 650,000 youth presented to the ED for violent injuries in 2008 alone. [62] In a national study of 4023 adolescents, 39% of teens with a history of assault (vs. 5% of teens with no trauma history) met criteria for major depressive disorder (MDD). [3] My pilot work shows that 40-60% of adolescents with a history of physical peer violence report past-month depressive symptoms, as compared to 17-20% of all teens seen in the ED. [9, 63-65] These rates are substantially higher than the 5-10% average 30-day prevalence of depressive symptoms in community samples of teens. [7, 66] Just as EDs screen for high-risk alcohol use or partner violence, a positive screen for past-year peer violence is a marker of being high risk for both MDD and future violent injury. [25, 67-72]

A strong theoretical basis exists to explain the bidirectional relationship between depression and violence. Many risk factors for depression—such as poor problem-solving skills, misreading of social cues, and inability to regulate one's emotional responses—also predict involvement in peer violence.[2, 13, 73] Depressive symptoms may therefore increase their risk of peer violence.[4, 5, 57, 74, 75] Conversely, peer violence may increase stress reactivity and reinforce maladaptive coping skills and negative world-views, thereby worsening depressive symptoms and potentially leading to MDD.[4, 10, 59, 69, 76-78] Targeted enhancement of cognitive and behavioral skills, to reduce both depressive symptoms and future peer violence, may be more effective for these high-risk adolescents.[28, 59, 79]

In sum, there is a strong bidirectional relationship between peer violence and depression in adolescents, due to common cognitive and behavioral errors. [1-4, 9] **This preventive intervention for adolescent ED** patients, uniquely tailored to reduce depressive symptoms in the context of peer violence, therefore has the potential to decrease depressed mood in the short-term within an extremely high-risk group.[34, 52, 80] If this research is successful, it could have a significant impact on the health of adolescents with minimal access to mental health services, high risk of developing more severe depressive disorders, and high rates of co-morbidities.

This K23 research plan therefore aligns with NIMH's Strategic Objective 3, to develop "new and better interventions for mental disorders that incorporate the diverse needs and circumstances of people with mental illness," and Objective 4, to "strengthen the public health impact of NIMH-supported research."

## (b) INNOVATION:

1: Development of an ED-initiated indicated depression prevention intervention for high-risk adolescents
Primary-care and school-based targeted CBT preventive interventions, some of which include elements of
motivational interviewing (MI) to increase participant engagement, are effective at reducing depressive
symptoms, mental health sequelae of violence (including PTSD), and psychosocial dysfunction.[28, 43, 81-85]
A single ED-based study using MI has been conducted (by Co-Mentor Cunningham), showing decreased
aggression among adolescents with both alcohol use and a history of peer violence.[42, 44, 86] Despite the
strong relationship between violence and depression, and the shared cognitive and behavioral deficits of these
disorders, no indicated depression prevention interventions exist for youth with a history of peer violence.

Adolescents with depressive symptoms and a history of peer violence often use the ED as their primary source of care.[31, 32, 87] They are unlikely to receive referrals to existing mental health services from the ED, unless they are seeking care specifically for psychiatric-related complaints.[8, 36, 63] Even when they do receive a referral, adolescents lack accessible mental health services.[30, 36, 88] Moreover, depression and violence are associated with low adherence to treatment.[89, 90] Therefore, while longer interventions may be more effective,[84, 91] *multi-session in-person interventions are unlikely to be successful with our population.*[89]

Brief ED-based interventions are effective at reducing recurrent suicidality and violence.[42, 44, 92-94] A brief, theory-based, ED-initiated depression preventive intervention for adolescents with a history of peer violence is therefore both indicated and innovative. The proposed intervention aims to decrease depressive symptomatology, and possibly prevent future violence-related episodes, in high-risk adolescents.

2: Use of state-of-the-art technology to improve reach, engagement, and outcome of this novel intervention.

Text messaging provides an ideal delivery mechanism to longitudinally engage and deliver content to these high-risk adolescents. Between 87% and 91% of teens, including those seen in the proposed study site ED,

own cellphones,[37, 64, 95] and adolescents average more than 50 text messages per day.[37] Theoretical benefits of a text-message-based longitudinal intervention protocol include continued engagement, real-life practice (e.g. daily text-message-based mood monitoring, goal-setting), increased dosage of therapeutic content, and the ability to tailor messages to participants' current emotional state.[41, 96-100]

Text-message-based interventions have been shown to be acceptable, feasible, and in some cases effective at delivering interventions addressing a variety of psychosocial issues, ranging from smoking to bipolar disorder.[38, 96, 101-103] A recent study in New Zealand showed acceptability, feasibility, and self-reported improvements in mood among adolescent participants in a school-based cell phone adaptation of a universal CBT depression prevention intervention.[39] Recent studies in American EDs showed that text-message-based alcohol[104] and diabetes[105] interventions are acceptable and feasible with young adult ED patients. No ED-based in-person or text-message interventions exist for reducing depressive symptoms.

Dr. Ranney (PI) has conducted surveys of the target population, showing their preferences for technology-based intervention formats,[64, 95] and is currently using text-messaging to assess adolescent girls' daily mood. Drs. Cunningham & Boyer have extensive experience developing technology-augmented interventions,[44, 106-110] although not for depression prevention. In this research project, Dr. Ranney will learn from her mentors' and advisors' previous research experience to develop an acceptable, single-session "ED" + longitudinal "text" depression prevention program for youth with a history of violence.

# (c)APPROACH:

**OVERVIEW OF PROJECT**: This project will develop, refine, and pilot a novel, single-session in-person + daily text-message ("ED+text") depression prevention intervention to reduce depressive symptoms among adolescents with a history of violence presenting to the ED for any reason. The intervention will target cognitive, affective, and behavioral strategies through a single, brief in-person introductory session ("ED") followed by 8 weeks of theoretically-informed text messages ("text") (**Table 11.2**). It is based on existing depression and violence prevention interventions as well as text-message preventive interventions developed for other populations.[38, 39, 104, 111]

The intervention has been designed, and will be tested, via an iterative process. In Aim 1 (ongoing, near completion) semi-structured interviews and expert consultation informed preliminary intervention content and format. In **Aim 2**, a series of small open trials and further qualitative analysis will refine it. In **Aim 3**, we

| Table 11.1: Inclusion/Exclusion Criteria for Screening | |
|---|---|
| Inclusion | Exclusion |
| ● Age 13-17 | <ul> <li>Acute suicidality/psychosis</li> </ul> |
| English-speaking | Sexual assault chief complaint |
| <ul> <li>Parent present and able to consent</li> </ul> | Child abuse chief complaint |
| <ul> <li>Medically/physically able to assent</li> </ul> | In police custody |

will then conduct a randomized, controlled pilot trial of the novel intervention among adolescents with depressive symptoms and a history of peer violence. We will use the same setting and participant screening/enrollment procedures throughout the study.

<u>Study Setting and Patient Population</u>: This study will be conducted in the pediatric ED of Rhode Island Hospital, which serves over 50,000 pediatric patients per year. The patient population is diverse, with 40% publicly insured, 40% Hispanic, and 25% African-American. Dr. Spirito has successfully conducted numerous studies of high-risk adolescents at this site.[47, 89, 112]

Patient Screening: The Research Assistant (RA) will be present on a random selection of shifts covering all days of the week, weighted by patient volume. Every patient meeting screening inclusion/exclusion criteria (see Table 11.1) who presents during an RA shift will be approached, in accordance with Dr. Cunningham's protocols. Only English-speakers (~95% of ED population) will be recruited for this development grant. Should Potentially eligible participants will be identified by RAs from the electronic ED tracking log. After obtaining parental consent/ adolescent assent, RAs will administer a computerized screen for depressive symptoms and past-year peer violence. The screen will also include basic demographic questions from the National Longitudinal Study of Adolescent Health (Add Health).[113] Additionally, to reflect my experience with 2 different screening processes during my pilot grant, we will administer some additional questions drawn from Add Health, YRBS, and other pertinent relevant measures of other behaviors (which I and my mentors have found increases participant honesty on all questions; in studies where we only administer the screening questions of interest, rates of self-report have decreased significantly). See Appendix 1 ("CODEBOOK") for questions.

Mentors Spirito and Cunningham have used similar screening protocols to recruit participant samples similar to the general ED population. All screened patients will be able to choose a small gift (\$1-\$2 in value) as compensation for their time.[86, 114]

<u>Eligibility and Enrollment</u>: Participants are eligible for <u>enrollment</u> if they screen positive for self-report of: (a) **depressive symptoms**, defined as a Patient Health Questionnaire-9 (PHQ-9)[115] score of  $\geq$  5, and b) **past-year peer (non-partner) violence** (victimization or perpetration), using a modified version of the Revised

Conflict Tactics Scale 2 [CTS2].[116] If meeting eligibility criteria, a second consent/assent and a detailed contact information form will be completed. If PHQ-9 score is > 20 or a positive answer to the suicidal ideation question, the attending emergency physician will be notified. Participants with severe depressive symptoms (PHQ-9 > 20) will be INELIGIBLE for participation in Aims 2 or 3. See Human Subjects for details. Refusal to permit audio-taping of ED sessions will be an additional exclusion criteria.

• Justification of eligibility criteria: (1) <u>Use of PHQ-9:</u> As per other depression prevention interventions, PHQ-9 is a standard screening tool to determine eligibility for targeted and indicated depression prevention studies.[43, 82, 83, 85, 117, 118] A cutoff of 5 accords with that used by other intervention studies.[119-121] (2) Adolescents reporting any past-

| Table 11.2: Theory-based Components of ED+text Intervention | | | |
|---|---|---|---|
| Theory/Model | Technique/strategy | Intervention Component | Delivery<br>Method |
| CBT, MI | Elicit recognition of problem(s) | -Feedback on depressive symptoms and peer violence - Identify "thought-feeling-action" triangle for negative thoughts & violence | In-ED +<br>Text |
| СВТ, МІ | Goal-setting | -Offer range of personal change goals for depression & violence, including option to create own goals - Separate personal goals from peer standards, particularly for violence -Convey respect & empathy for goals - Define "rewards" for meeting goals | In- ED +<br>Text |
| СВТ | Cognitive restructuring: - Challenge negative thoughts - Problem-solving | - Identify negative thoughts, their triggers, and their results (emphasizing violence's role as trigger/outcome) - Identify alternatives to negative thoughts and violence - Encourage non-violent assertiveness - Put negative events in perspective | Text |
| СВТ | Affect regulation: - Emotional regulation - Distress tolerance | Identify alternative ways of dealing with common stressors and potential fights ("coping plans") Provide strategies to calm down and deal with stress and threats | Text |
| СВТ | Behavioral<br>activation: | - Develop a list of fun, non-violent activities (social, physical, and indulgent) - Elicit pro-social behavioral skills - Reminders of community mental health/violence-prevention resources | Text |

<u>year peer physical violence</u>. "Peer" violence is non-partner, non-family-perpetrated physical violence. Adolescent peer victimization and perpetration strongly overlap, and teens with *any* past-year fights (not just those with acute injury) are high risk for future injury and depressive symptoms.[3, 122] Co-Mentor Cunningham has used the modified version of CTS2 for multiple ED-based studies addressing peer violence.[44, 86, 113, 116, 117]

• Justification of enrollment feasibility: Each month ~1200 patients age 13-17 present to the RIH ED. Based on AIM 1 results, approximately 20% of teens will screen positive for both current depressive symptoms and past-year peer violence; in Aim 1, 70% of eligible teens consented for interviews. At a very conservative 50% consent rate, at least one participant would consent per eight hour recruiting shift (~20 pts/month). High retention rates (~80%) are reported by her mentors and others in similar longitudinal intervention studies.[39, 42, 47, 96, 104] See Figure 11.1 (under Aim 3) for flow chart.

#### AIM 2: Refine intervention content:

In this Aim, the newly developed depression prevention intervention will be iteratively refined, recruiting four adolescents per round (two of each gender) for at least four rounds of open pilot testing (a total of at least 16 adolescents). Under the guidance of her entire mentorship team, Dr. Ranney will use semi-structured interviews and measures of protocol adherence to evaluate and then improve the intervention's appropriateness and comprehensibility for the target population. The open trials will also provide an opportunity to assess the feasibility of inclusion and exclusion criteria, and recruitment and assessment procedures.

• <u>Study setting, eligibility, and enrollment</u> are as above. Additionally, participants will need to own or have access to a cellphone that can receive text messages. A subset of the participants in Aim 1 (who have previously consented to be contacted) will be contacted via mail and cellphone to see if they want to participate in Aim 2. We will limit cross-enrollment to a maximum of 1/3 of our sample.

Open trials will last for the full anticipated intervention duration of 8 weeks.

- <u>Incentives</u>: \$25 for completing the baseline assessment and in-ED intervention, \$10/month for text-messaging plans, \$5 for completing follow-up survey prior to the follow-up interview and \$50 at follow-up interview.
- "ED" session (~20-30 minutes): This session will take place during waiting periods in the ED stay; average ED visits are 3-5 hours. The session is a manualized adaptation of the first session of an effective CBT-based depression prevention program (provided to the PI by Dr. Paul Rohde, who is available to advise on an as-needed basis)[43, 82] and of Cunningham's MI-based violence interventions.[44] Using Spirito's and Cunningham's brief ED interventions as a model, the trained interventionist will provide participants with immediate feedback, using computerized baseline assessment scores (a very brief version of the planned baseline assessment, to help us refine the intervention). The interventionist will then give a brief overview of Beck's Cognitive Triad (the interplay between thoughts-emotions-behavior); and will conduct personalized goal-setting using MI techniques (Appendix 2, "ED SESSION"). Participants will also be oriented to the text-message system, including potential human subjects concerns (see **Human Subjects**).

During the session, the parents will be asked to step out of the room. They will be given publicly-available content regarding adolescent depression prevention to review, both to enhance their buy-in to the project and to occupy them during the intervention.

All sessions will be audio taped. Following each session, the interventionist will complete an adherence rating form to indicate how well the protocol was followed. Adherence manuals will be developed by Dr. Ranney and Spirito based on session content, the Cognitive Therapy Rating Scale (CTRS),[49] and the Motivational Interviewing Treatment Integrity Code (MITI),[50] well-validated methods of assessing competence and adherence. **Mentor Spirito will listen to all sessions with Dr. Ranney as a training activity**, and as part of the treatment development process. After each round of open pilot testing (4 participants each), the "ED" protocol will be modified according to participant and interventionist feedback.

• "<u>Text" component (daily for 8 weeks):</u> Based on results from Aim 1, we will sending *one automated assessment followed by one tailored CBT-informed text message each day*, at a time of the participant's choice. Each week, a variety of messages will be delivered to create both (a) a natural progression in skill-building; (b) continued motivation for participation; and (c) responsiveness to participants' needs, through tailoring. This daily text-message system will maximize active engagement and increase participants' practice of key CBT-based concepts, which has been shown to correlate with change in depressive symptoms.[84] We will also provide *participant-driven text-messages*: e.g., if the participant texts "FIGHT" or "MOOD" to the

automated program, indicating need for additional support on that topic, s/he would receive an appropriate skill-based message.

After each round of open testing, message prompts, content, and frequency will be **iteratively refined based on qualitative and quantitative assessments**. Final content will be submitted to the IRB prior to the start of Aim 3 (at which point the intervention will not be further revised). The current conception of the messages and the delivery algorithm are attached as **Appendix 3** ("TEXT MESSAGES").

Messages will be delivered to participants' own cell phones using an automated computerized system developed by an outside company, Reify Health, based on pre-specified delivery algorithms. Any responses that deviate from expected requests will receive an automated "crisis message." Data from the responses will be reviewed weekly, and will be visible ONLY to members of the research team (see **Human Subjects**). (see **Appendix 3** and **Human Subjects** below).

PI Ranney used this system to conduct daily mood assessments of high-risk adolescent girls in a pilot grant funded by a private foundation with over 80% response rates to 9 daily

messages and overwhelmingly positive feedback during a post-assessment interview. Mentor Spirito is currently using Reify Health to deliver text-messages for an NIMH-funded R34 for adolescent suicide prevention. Advisor Boyer has successfully delivered interventions to participants using a similar system.

• <u>Assessments:</u> In addition to the assessments in the screening protocol, we will administer assessments at the close of the open intervention to guide refinement of the "ED+text" intervention. Specifically, we will



collect data on feasibility: study recruitment and refusal rates, program completion, follow-up rates, reliability and range of responses to baseline and follow-up questionnaires, and rates of study attrition (see CODEBOOK AIM 2). Participants will also complete detailed qualitative debriefing after the in-person and text-messaging components of the intervention (see QUALITATIVE ASSESSMENT). This evaluation necessarily occurs on a clinical, non-statistical level. Participant acceptance of the text-messaging will also be assessed by: (1) The System Usability Scale, a participant-completed, reliable and valid metric for measuring usability and acceptability of technologies.[123, 124] Higher scores equate to higher usability.[125, 126] (2) Relative Subjective Count (RSC), the quotient of the participant's estimate of the number of times the system delivers a text, divided by the actual number of texts delivered.[127, 128] As text-message systems are unable to track actual number of texts opened, this measure is a reliable surrogate measure of acceptability.[127, 128] Low RSC (e.g., <1.0) correlates with increased participant satisfaction, while elevated RSC (>1.0) reflects poor acceptability of a technology (e.g. that the messages were intrusive).[127, 128] Lastly, in recognition of the NIH's move toward "learning healthcare system" outcomes, we will include a review of Lifespan electronic medical records (EMR) to determine participants' ED visits and admissions over the 8 weeks of the study period, to show the feasibility of tracking this data. We will extract only the number, category, and disposition of the visits (specifically, whether the visit was related to injury, psychiatric complaints, or medical complaints, and whether the patient was discharged, transferred [as well as transfer location], or admitted to Hasbro) from the Lifespan EMR.

# Aim 3: Conduct a pilot randomized trial of the novel "ED+text" intervention versus enhanced usual care (EUC).

This Aim corresponds to **Stage 1b of intervention development (pilot testing and refining the intervention)**.[129] In Years 3-5, a two-group randomized design will be used to measure intervention feasibility (numbers of patients recruited, retained, randomized, and completing all follow-ups) and acceptability (satisfaction questionnaires and exit interviews), as well as exploratory hypothesis testing. In Year 5, analysis and grant authorship will occur. The entire mentorship team will guide Dr. Ranney in this Aim.

- <u>Intervention Recruitment:</u> Participant screening and enrollment processes will remain the same. Study setting, eligibility, and enrollment are as per above, with the additional requirement (as per Aim 2) that participants own or have access to a cellphone that can receive text messages.
  - Content: Per above.

• <u>Study Randomization and Intervention Conditions</u>: Eligible participants will be randomized to experimental (ED+text, n=50) or enhanced usual care (EUC, n=50) care. As gender is a known moderator of depressive symptoms and violence, [12, 58, 73, 136] randomization will be stratified by gender and baseline depressive symptoms, using block randomization. See **Figure 11.1** for flowchart. All participants will complete

a baseline assessment in the ED. If randomized to ED+text, they will complete the introductory session during waiting periods in their ED visit (as per Drs. Spirito's & Cunningham's ED-based interventions), then will receive daily tailored CBT-based textmessages for 8 weeks. EUC will consist of a brief introduction to home safety and nutrition, as well as an introduction to the text-message service in the ED, followed by eight weeks of regular text messages on safety, diet and nutrition. The current standard of care for these patients is, in essence, no care: no depression or violence screening assessment protocols are currently used in our ED. Both "ED+text" and EUC conditions therefore exceed current levels of care.

| Table 11.3: Schedule of Participant Assessments | | | | |
|---|---|---|---|---|
| Construct | Measures | Baseline | 8-<br>week | 16-<br>week |
| Depressive symptoms | BDI-II[130, 131] | Х | Х | Х |
| Peer violence | CTS-2 (physical<br>subset)[116]<br>YRBS Physical Fight | х | X<br>X | X<br>X |
| | CADRI (physical subset)[132] | | Х | X |
| Cognitive/behavioral skills | IPAS Positive Affect Violence Self Efficacy Short Hopelessness Scale Emotional Regulation Rumination | X<br>X<br>X | X<br>X<br>X<br>X<br>X | X<br>X<br>X<br>X |
| Associated co-<br>morbidities | Substance Use Child PTSD Symptom Scale[134] | X | Х | X |
| Resource utilization | Child & Adolescent<br>Services Assessment[135] | | | Х |
| Process measures | Client Satisfaction Questionnaire-8[48] | | Х | |
| | Relative Subjective Count | | X | |
| | Qualitative assessment | | X | |

• <u>Assessments</u>: At screening participants will be asked additional questions from the Child & Adolescent Services Assessment, the Short

Hopelessness Scale. Other question types include: medication use, delinquency, drug use and binge drinking, community violence, intimate partner violence (CADRI physical subset), symptoms of Post-Traumatic Stress Disorder (PTSD), safety and nutrition factors, cell phone use, cyberbullying, access to medical services, and demographics. These will be in addition to screening eligibility questions (CTS-II and PHQ-9).

We will assess depressive symptoms, violence, cognitive/behavioral skill-sets, and resource utilization at baseline; 8 weeks (at the close of the text-messaging portion of the study); and 16 weeks. Although a longer follow-up period would be preferred, these follow-ups were chosen based on budgetary and time constraints of this training grant. In accord with mentors' ED studies,[42, 47] assessments are expected to take ~30 minutes to complete. They have been modified based on Aim 2 data. Although limited in the baseline assessment due to in-ED time constraints, we recognize that a number of important co-morbidities, such as substance use and PTSD, may relate to our intervention's effectiveness. We will measure these at screening, baseline and follow-up. At the 8-week follow-up, standardized quantitative process measures will be administered to assess acceptability, usability, and feasibility; qualitative interviews will be administered to a purposefully sampled subset of a maximum of half of both the intervention and control groups.[124, 137] (See Table 11.3 and Appendix F for details on assessment schedule and psychometric properties). Lastly, in recognition of the NIH's move toward "learning healthcare system" outcomes, we will include a record of maximum heart rate during the ED visit, and review of the EMR for ED visits and admissions over the 6 months following enrollment in the study, as described in the Aim 2 protocol above.

- <u>Fidelity Protocol</u>: The fidelity of the text-message component is assured, as all text-messages will be automated. To assess fidelity of in-person ED sessions, all will be audio-taped. The interventionist's first 10 tapes will be rated by Drs. Spirito and Ranney, *according to guidelines to be developed in Aim 2*, to objectively evaluate if there is protocol drift. If tapes meet the 80% criterion, 20% of recordings thereafter will be coded. Criteria for adherence to the ED session will be defined in terms of specific content areas, as well as adherence to basic CBT and MI principles.[49-51] **This will serve as a training activity.**
- <u>Incentives:</u> Maximum compensation for completion of the entire trial will be \$150 (\$25 for baseline, \$40 for 8-week follow-up, \$50 for 16-week follow-up, \$20 for unlimited text-messaging plan for 8 weeks, \$5 for alerting us to a change in phone number, \$5 each for finishing the 8 & 16 week follow-ups online). Spirito and Cunningham have successfully recruited and retained 80-90% of participants for 12-month follow up across multiple trials with high-risk adolescent ED patients, using similar protocols and compensation.[42, 47, 89]

Mental Health Safeguards and Data Management: The research assistants will be extensively trained by the PI and Mentor Spirito to recognize and manage participant distress. In case of severe depressive symptoms, suicidality, or other crises during in-ED screening, the interventionist will immediately notify the PI and the attending emergency physician. If mental health crises are identified during interviews outside the ED, the research team will contact the PI at time of identification and refer appropriately, according to the drafted crisis plan. Mentor Spirito, a licensed clinical psychologist, will be available by phone for clinical decision-making. Please see **Human Subjects** for further details.

#### STATISTICAL ANALYSIS

<u>PHASE ONE, Aim 2</u>: Using data collected during the open trials, we will perform a <u>preliminary process</u> <u>analysis</u>, examining study recruitment and refusal rates, study completion rates, use of text messages, follow-up rates, reliability and range of responses to assessments, and overall study attrition. We will study exit interview transcripts for acceptability, treatment satisfaction, and comprehensibility. Exit interviews will also undergo <u>thematic analysis</u>, similar in methodology to Aim 1. Because the interview topics are restricted to review of the revised materials and feedback on planned intervention components, it is likely that most codes will be deductive. Analysis will also focus on key domains that are also covered by the quantitative evaluation instruments so that the qualitative data can provide additional context for that quantitative data.

In addition, as described in Aim 2: Assessments, above, we will assess the text-messages' usability and acceptability by calculating the mean score for the <a href="System Usability Scale">System Usability Scale</a> (SUS)[124, 125] and the <a href="Relative Subjective Count">Relative Subjective Count</a> (RSC).[127, 128] The SUS will be administered at the close of the 8-week intervention; a higher score correlates with higher usability. The RSC will be calculated based on information obtained in the exit interviews, as successfully used by Dr. Boyer; lower scores correspond to higher acceptability.[127, 128] We will also review the number and type of ED visits and hospital admissions for the duration of the study to examine trends in hospital admission as an effect of study participation.

Based on these formative data, we will further refine our intervention and study protocol.

### PHASE TWO, Aim 3:

- <u>Sample size</u>: For this intervention pilot study, we chose to recruit 120 subjects in the RCT. Conservatively estimating that 20% may be lost to follow-up, 96 subjects will complete the 16-week assessment. This number will be sufficient to allow us to make judgments regarding feasibility and acceptability. Despite problems in the stability of effect size calculations with small samples, if a small effect size is detected between groups, and the intervention is shown to be feasible and acceptable, then further testing in a larger trial may be indicated given the innovative nature of the intervention and its potential disseminability.[138, 139] Based on our Aim 1 results, we anticipate that the mean PHQ-9 score of our participants will be 10.0, with a standard deviation of 4.5. If we wish to show a delta-PHQ9 of 2 (with alpha 0.05 and beta 0.8), we would need to successfully follow up 63 participants.
- <u>Data management:</u> Data from text messaging, including time of delivery and any participant responses, will be stored in a de-identified database on a HIPAA-compliant server. This de-identified data will be imported into Stata 12 (Stata Corp, College Park, TX), with which I and my mentors are skilled. Stata 12 is suitable for the multi-level modeling necessary for a fully-powered longitudinal study.
- Acceptability and feasibility (Aim 3a): Acceptability will be measured using descriptive analysis of enrollment rates, participants' ratings of the clarity and structure of the in-person and text-message sessions, Client Satisfaction Questionnaire-8,[48] Feasibility will be measured using percent of in-person sessions completed, the RSC (as described in Aim 2).[127, 128] and therapist adherence ratings.
- Exploratory hypothesis testing: We will calculate total scores for depressive symptoms (PHQ-9, BDI-II) and violence exposures (CTS-2, CADRI) at baseline and follow-up. We will calculate descriptive statistics for study sample demographics, baseline mediators/moderators (e.g. IPAS, hopelessness), co-morbidities (CPSS) and service utilization (CASA). T-test and chi-square comparisons will be used to detect baseline between-group differences.

The *primary exploratory outcome* of interest is depressive symptoms (measured by BDI-II); the *secondary outcome* is peer violence (CTS-2). Under Dr. Papandonatos' guidance, we will first calculate preliminary estimates of the between-groups differences in depressive symptoms (continuous) and peer violence (counts), with 95% confidence intervals, at 8- and 16-week follow-up assessments, adjusted for baseline values. An intent-to-treat approach (all patients randomized to intervention will be retained in analysis) will be used to address potential problems inherent in following only treatment completers and the potential for differential attrition across conditions.[140, 141] In cases of loss-to-follow-up, baseline observations will be carried forward.

Generalized linear mixed models (GLMM)[142, 143] that employ likelihood-based estimation approaches will then be used to evaluate changes in depressive symptoms and number of fight episodes at the 8-week and 16-week follow-ups. Intervention condition will be considered the primary predictor variable. Race and gender will be included as secondary predictors. We will control for baseline levels of the outcome variable (e.g. severity of baseline depressive symptoms and peer violence) as well as the linear and quadratic effects of time. We will also examine potential moderators of the intervention effect, including gender, race, and baseline coping skills. In GLMM, no missing data imputation will be employed, as the models produce consistent estimates in the presence of data missing-at-random.[144, 145] **Analyses will serve as a training activity.** 

Potential Problems & Alternative Strategies: Parental involvement: According to pilot data, 99% of eligible adolescents seen in our ED are accompanied by a parent. We recognize the importance of parents in teens' mental health, but we have chosen not to include parents any further than the consent process, in order to focus on acceptability for adolescents, [146] and to increase feasibility and eventual disseminability. Difficulty completing in-person session during time in ED: My mentorship team has successfully completed multiple studies with 45-60 minute CBT- and MI-based interventions for teens in the ED. Enrollment biases: Patients who are more symptomatic or more comfortable with technology may be more likely to enroll. In our planned R01 we will correct for these characteristics by stratifying by baseline symptom severity, and by including technology use as a covariate; we will also adapt the intervention for Spanish speakers. Attrition of participants: Our study recruitment location has a strong track record in retaining our target population in longterm studies. I will conduct weekly meetings with staff to identify potential threats to participant retention. The native attraction of text-messaging to adolescents should help prevent fatigue from intervention use [39, 147, 148] Although we anticipate 15-20% attrition based on past work, we believe that we can respond rapidly and effectively to any potential difficulties. Technology difficulties: Through the PI's foundation grant and Dr. Spirito's NIMH-funded R34, we have successfully piloted the text-message technology that we propose to use in this project. Cell phone concerns: Participants will be compensated for their monthly text-messaging plans. See **Human Subjects** for details on protection of confidential information, and for mechanism to regain contact in case of changed phone numbers.

#### 14. PROTECTION OF HUMAN SUBJECTS

<u>Summary</u>: For this clinical study, all data collection sheets and computerized databases will use a unique numeric code to identify specific subjects. The code sheet will be kept in a locked file cabinet in Dr. Ranney's locked office, and on password protected files on secure hard drives owned by Dr. Ranney's institution. We intend to seek approval for this study from the human protection committees at Rhode Island Hospital; no study activities will be initiated without full institutional review board approval. All members of the research team have already completed training and received certification in Human Subjects Research Protection (CITI Program) and HIPAA regulations. They will continue to renew this training in compliance with Rhode Island Hospital and Brown University policies. Additionally, a **Certificate of Confidentiality will be obtained** for this study from NIH once IRB approval has been granted.

### 14a. Risks to the Subjects

## 14a.1. Human Subjects Involvement and Characteristics:

In Specific Aim 2, approximately 16 adolescents will participate in a series of open trials of the ED-based preventive intervention. In Specific Aim 3, the novel "ED+text" intervention will be studied in a randomized controlled pilot trial, with 50 participants in the "ED+text" arm and 50 participants in the enhanced usual care (EUC) arm. The ethnic and racial composition of the study group will be expected to represent that of the pediatric population seen in the Rhode Island Hospital ED, identified to be approximately 40% Hispanic and 25% black or African American by my own pilot study (data analysis in progress). Children aged 13 to 17 will be included in the study.

Inclusion Criteria. To recap what was described in Section 11c above: Inclusion criteria for screening include: being medically stable; mentally and physically able to assent; English-speaking; and having a parent present to consent. Exclusion criteria for screening include a chief complaint of sexual assault or child abuse; a chief complaint of acute suicidality or psychosis; or being in police custody. Additional inclusion criteria for enrollment (in Aim 2 or Aim 3) include a PHQ-9 score > 5 and past-year peer violence (according to CTS2).

Potentially eligible participants will be **excluded** from enrollment if they or their parents do not consent to audio-taping of the in-ED session or if they meet criteria for severe depression (PHQ-9 > 20). Additionally, patients who are deemed (based on in-ED assessment by a clinician, after notification about a positive screen for suicidality) to need a psychiatric hospitalization will be ineligible.

Participants in Aim 1 may be eligible for Aim 2, but will be restricted to less than 1/3 of the Aim 2 sample. Participants will be ineligible for Aim 3 if they have participated in Aims 1 or 2.

Rationale for including special classes of subjects. This research will involve children between the ages of 13 and 17 inclusive. The age range is dictated by the prior research showing elevated risk for depression and peer violence among teens in this age range. It is of utmost importance to study this "vulnerable population" because they are an understudied population; a population at high risk of negative outcomes; a population with limited access to and use of traditional mental health services; and a population with high possible benefits if effective, accessible preventive services can be developed.

All ethnicities and races will be equitably included. Only English-speaking patients will be eligible for two reasons. First, our previous and ongoing studies show that the vast majority of Hispanic adolescents speak fluent English.[9, 149, 150] Second, due to budgetary constraints inherent in this training grant, it would be difficult to fund a bilingual interventionist and translation of all materials into Spanish.

#### 14a.2. Sources of Materials:

Materials will be collected from adolescent participants in the study. Data will be collected from participants primarily using a tablet laptop computer and audio-taped interviews; some de-identified data may be collected through secure text messaging services in Aims 2 and 3. Minimal data will be collected from Medhost and Lifelinks regarding participants' ED utilization and hospital admissions after initiation of the study. Data that are obtained specifically for research purposes will be collected only with written assent from youth and written consent from a parent or guardian. Minimal clinical data will be collected on patients that refuse to participate in the study, on patients that the research assistants fail to approach about the study, and on patients that are excluded from the study. This data will be obtained from de-identified emergency department medical records, to assess characteristics of patients not approached or who refuse participation.

<u>Linkages to subjects and access to subject identities</u>. For each stage of the research, participant names and contact information will be maintained in a secure, password-protected recruitment/enrollment database. Once individuals enroll in the study, names will be linked to participant ID number *only* in this database, which will be kept in a restricted access folder on a secure server. This file will be assigned a code name unrelated

to the name of the study. Baseline, follow-up, and focus group data will be coded according to participant ID number, and will contain no protected health information.

To facilitate scheduling the 8 week follow-up interview during Aim 2 only, participants *may* choose to participate in the YouCanBookMe Limited scheduling service. This is a voluntary third party, encrypted service that schedules appointments using the participant's email address, first initial, and last initial. The data will only be scanned by the system for the purposes of scheduling and rescheduling the participant's follow-up interview. Once the scheduled interview is complete, members of the research team will erase the participant's email from the YouCanBookMe encrypted server. While this information will be kept in confidence by the research team, and while YouCanBookMe assures that it will not access the information for any promotional purpose, we cannot prevent outside forced entrance into the YouCanBookMe server.

Signed consent and assent forms will be kept in a double-locked file cabinet in the PI's locked office, separate from any other project data. Once data collection for each stage of the study is completed, the corresponding recruitment/enrollment database will be deleted as it is unnecessary to maintain the link between participant identity and study data. All information collected as part of this study will be accessible only to research staff that has completed mandatory training in the protection of human subjects.

<u>Data collection</u>. Data will be collected solely for the purposes of this research project. All information collected as part of this study will be obtained only by research staff employed by the project. Data sources include: 1) participants' responses to baseline and follow-up questionnaires, 2) confidential audio-taped semi-structured interviews, and 3) participants' responses to text-messages. In Aim 2, data will be collected at screening, baseline and after the intervention. In Aim 3, data will be collected at screening, baseline, 8 weeks post-enrollment, and 16 weeks post-enrollment.

#### 14a.3. Potential Risks:

Every effort will be made to ensure that study participants are protected from risks. The risks are as follows: 1) potential coercion, 2) loss of confidentiality, 3) emotional discomfort during the assessment and/or program sessions, and 4) further violence if an assailant is made aware of program involvement. The protection against each risk is described in detail in **Section 14b.2**, **below**.

## 14b. Adequacy of Protection Against Risks

# 14b.1. Recruitment and Informed Consent:

Screening and Consent. A research assistant (RA) will be present in Hasbro Children's ED on randomly selected shifts (selection weighted according to patient volume). All patients between ages 13 and 17 will be pre-screened by the RA. If the patient is triaged as stable, and is not presenting for with a chief complaint of suicidality, psychosis, sexual assault, or child abuse, the RA will approach the patient and his/her family once the patient is put in a private treatment room. After reading a script to the parent and child, verbal consent/assent will be obtained from the parent/legal guardian and the child. Then, youth will complete a computerized screening survey. The adolescent and his/her parent will be informed that the adolescent's answers to study questions may be used to determine their eligibility for a research program. After completion of assent/consent, the teen will then be administered the screening questionnaire, including PHQ-9, and CTS-2. Additionally, to reflect my experience with 2 different screening processes during my pilot grant, we will administer additional questions drawn from Add Health, YRBS, and other relevant materials about other behaviors (which I and my mentors have found increases participant honesty on all questions; in studies where we only administer the screening questions of interest, rates of self-report have decreased significantly). All participants will be able to choose a small gift (worth \$1-2) as compensation for their time.

If an adolescent screens positive for mild-to-moderate depressive symptoms (PHQ-9 between 5 and 20) and past-year peer violence, s/he will be informed that they are eligible for the research program. Adolescents and their parents will be informed that their responses to screening questionnaire indicate that they are eligible for a program to help build mental health and prevent fights. Screened participants who agree to be part of the study will complete an additional *written* assent/consent form for Aims 2 and 3.

All individuals who agree to participate in the screening will be given referral information for a variety of community resources including community mental health services and violence prevention organizations.

During recruitment, research staff will inform the subject of the general nature of the study, their privacy rights, expectations for their participation, the voluntary nature of their participation, and that their participation can be withdrawn at any time. Participants will be assured that refusal to participate will not affect their care in any way. At all times, research staff will make explicit the voluntary nature of the subjects' participation as well as potential situations for breaking confidentiality. Recruitment procedures will be HIPAA compliant and have been IRB approved in past studies.

<u>Referrals.</u> All participants in the screening will receive a handout of mental health and violence prevention resources. If an adolescent screens positive for severe depressive symptoms at any time during the study, regardless of eligibility for the study, the RA will discuss the score with the family, notify the attending pediatric emergency physician, and offer to contact the adolescent's pediatrician.

If an adolescent discloses suicidality or if the patient's family so desires, the RA will alert the patient's clinician (if appropriate) who will immediately initiate a psychiatric evaluation in the ED, or will contact the patient and his/her parent if disclosure occurs outside of the ED. (See "Mandatory Reporting & Crisis Management," below). If a patient is deemed to need psychiatric hospitalization based on the screening, they will be withdrawn from the study.

Assessments and Remuneration. In **Aim 2**, participants will complete a baseline assessment, an 8-week follow-up assessment and interview; **in Aim 3**, participants will complete a baseline assessment, an 8-week interview and an 8-week and 16-week computerized follow-up assessment. Follow-up assessments will take place online, on the telephone, or in private rooms at the PI's departmental office (separate from the ED) where privacy and confidentiality can be maintained (i.e., making sure no one can overhear the conversation).

Participants will be remunerated with a gift worth ~\$1-2 for the screening survey. In **Aim 2**, participants will be compensated \$25 after completing the baseline assessment and in-ED intervention, \$10/month for text-messaging plans, an additional \$5 incentive if they complete the 8-week follow-up survey *prior* to the 8-week follow-up interview, and \$50 for completing the 8-week follow-up. In **Aim 3**, participants will be remunerated \$25 after completing the baseline assessment and in-ED intervention, \$40 for completing the 8-week follow-up, \$50 for 16-week follow-up, and \$10/month for text-messaging plans. Participants will also receive \$5.00 for notifying us of any address/telephone changes, and an additional \$5 for completing the 8-week and 16-week surveys *prior* to their due date.

# 14b.2. Protection Against Risk

# Risk 1): Potential Coercion.

The risk of potential coercion will be minimized by following standard procedures for obtaining the informed consent from parents and assent from teens. Study personnel will fully explain the study procedures, risks, benefits, and alternatives to teens and their parents. Participants and their parents will also be reminded that study participation is voluntary and that refusing to participate or withdrawing from the study at any time will not result in any negative consequences on their care.

### Risk 2): Confidentiality

Potential risk will be minimized by strictly adhering to the guidelines for research outlined by the Lifespan IRB, Rhode Island state law, the Federal Health Insurance Portability and Accountability Act of 1996 and its regulations ("HIPAA"), and the DHHS Federal Policy for the Protection of Human Subjects (45 CFR Part 46 Subpart D). In particular, the risk of loss of confidentiality will be minimized by the following specific procedures:

## **UNIVERSAL:**

- (a) All research staff will sign a pledge of confidentiality and will understand that violation of confidentiality is reason for dismissal. Training of staff includes information about the importance of confidentiality and techniques to maintain confidentiality of all information reported by research participants.
- (b) Any collected information will be referenced only by participant ID #.
- (c) The only list connecting the participant ID # to the participants' names will be kept in a password-protected folder on the PI's password-protected computer (which is owned by the hospital, and which is on the hospital's HIPAA-secured research server). This list will be deleted as soon as each phase of the study is completed.
- (d) The consent forms and research materials will be kept in separate double-locked cabinets in the PI's locked office.
- (e) All computerized information will be maintained on password protected, HIPAA-compliant computers owned by the PI's hospital which use only HIPAA-compliant research server.
- (f) All computerized surveys will be completed using REDCAP.
- (g) No names, only identification codes, will be used in presenting data in lectures, seminars, and papers.

# **SEMI-STRUCTURED INTERVIEWS:**

(a Semi-structured interviews will take place in a private room at the site of the participant's choosing (e.g. ED, Pl's departmental office, library, telephone) where confidentiality can be assured

- (b) Ground rules will be set at the beginning of the interviews, instructing participants to not identify themselves or others by name, and emphasizing the confidentiality of everything discussed [with the exception of suicidality/homicidality/child abuse].
- (c) Participants will be not be referred to by name on the audiotapes.
- (d) Prior to transcription, the digital tapes will be kept in a password protected format on a password-protected Lifespan hard-drive accessible only to the PI and the RA. The recordings will be maintained for 5 years in compliance with human subjects policies.
- (f) Transcripts will be reviewed only by the PI and her research team.

# TEXT-MESSAGING:

- (a) All text-messages will be sent using a secure text messaging system (hosted by Reify Health, a company that we have worked with in the past for similar projects) that will not store data remotely; the text-message server is located behind a research-compliant firewall.
- (b) Text-message data will be maintained in a password-protected, restricted-access hard drive in the Department of Emergency Medicine.
- (c) Text-message data will be monitored exclusively by the PI and her research team.

Participant confidentiality will be breached only to protect the safety and welfare of research participants and only in accordance with state and federal law. The exceptions to confidentiality include if the adolescent reports suicidality, homicidal thoughts, or that he/she is the victim of child abuse or neglect. If the adolescent reports suicidality or homicidality, parents will be notified, and an emergency psychiatric evaluation for inpatient hospitalization will be facilitated with the Pediatric Emergency Psychiatric Service at Rhode Island Hospital. If necessary, authorities will be notified. If child abuse or neglect is reported, a report will immediately be filed with the Department of Children, Youth and Families. This exception to breaking confidentiality – the case where a participant reveals child abuse, suicidality, or homicidality – will be explained in detail to both participants and parents prior to completing the assent/consent.

Finally, information collected in this research study will not be available to clinicians, parents, or to other researchers. All data will be collected specifically for use on this project.

# **Risk 3) Emotional Discomfort**

Of note, members of the proposed mentorship team have substantial prior clinical and research experience with high-risk populations as evidenced through their biographical sketches. Dr. Spirito has extensive clinical and research experience developing interventions for depressed, suicidal, and alcoholabusing adolescents. Dr. Cunningham has extensive clinical and research experience with adolescent violence and substance abuse prevention.

<u>Parental distress:</u> If parents report feelings of distress as a result of being notified that their child is eligible for this research project, clinical resources will be offered. These include referrals for mental health counseling and information about violence hotlines and local community organizations.

<u>Assessments:</u> The assessment instruments are commonly used in research and clinical practice. We will minimize distress by presenting questions/program techniques in a supportive manner, assuring participants that they may refuse to answer questions that make them uncomfortable, and reminding them that they may terminate the assessment and/or intervention at any time.

Although there is extremely low risk of an adverse reaction to the screening survey or qualitative interviews (and, in fact, benefits to participation in similar research have been demonstrated),[151] all potential participants will be provided with a list of community resources at the same time that they are approached by the RA about participation in the study. To minimize negative consequences from the screening survey or semi-structured interviews, the RA will be trained to immediately terminate the assessment and alert the PI and the patient's clinician in the case that the subject demonstrates physical or psychological instability.

Additionally, on completion of baseline and follow-up assessments, the RA will be alerted by the computer if a participant has reported suicidality or severe depressive symptoms. The RA will contact Dr. Ranney or Dr. Spirito at that time, and the teen will be further evaluated for risk of harm to self or others. To the extent that the adolescent is determined to be a risk to himself/herself or others, the parent will be notified and a referral to an emergency evaluation with the Pediatric Emergency Psychiatric Service at Rhode Island Hospital will be made.

Regarding the text-messaging component of the study, text message assessments do NOT induce depression despite repeated assessments of negative mood.[152] Momentary assessments have also been shown to be acceptable, feasible, and appropriate when used to ask sensitive assessments (e.g., suicidality,

mood, alcohol and substance use, eating disorders, and violence) among a variety of populations, including school-age adolescents, schizophrenics, the homeless, drug addicts, recently hospitalized suicidal patients, and college students.[153-163]

<u>Text-message Data:</u> Participants and parents will be explicitly instructed during the consent process that no one will be monitoring text-message data in real time. In the case of a crisis situation, the adolescent should call the provided crisis hotline number or the Pl's phone number rather than text the program. Nonetheless, some participants may misinterpret these guidelines. Hence, text-message data will be reviewed regularly by the Pl and her mentorship team. <u>The software will also be designed to send participants a message that directs them to a crisis phone number, if data that is not expected by the text-message algorithm is received.</u>

OF NOTE: This protocol mirrors that used by other text-message-based interventions for mental health and other potentially sensitive behaviors/disorders (e.g. [39, 104, 164-168]), including one that is currently ongoing with Dr. Spirito and Dr. Ranney at Brown University (for suicidal adolescents). Moreover, as the text messages include \*no\* PHI and \*no\* sensitive information regarding diagnoses, they easily meet or exceed HIPAA regulatory standards [169].

Ongoing Safeguards: Due to the association between violence and mental health sequelae, it is possible that some participants will experience psychiatric symptoms during the course of the program that may warrant mental health care. In order to minimize the risk of mental health deterioration, all subjects may receive mental health treatment at any time during the study. Clinical need will determine whether it is appropriate for the participant to continue in the study.

The PI's email and phone number, and a crisis hotline number, will be provided to every participant. The participant will be instructed to call the PI in case of any problems with the study, or if s/he has an immediate mental health crisis. S/he will be encouraged to call the crisis number, or 911, as well, if in need of immediate mental health services. The participant will also be provided with a wallet card explaining why she is responding to text messages, in case s/he is asked by a teacher or employer.

If a participant is identified as needing mental health treatment, the PI or her mentors will contact the participant individually for further assessment, and will notify the participants' parents of any clinical needs. Evaluation by the Pediatric Emergency Psychiatric Service at Rhode Island Hospital will be initiated on the PI's discretion at any sign of suicidality, homicidality, or child abuse. Suicidal or homicidal attempts or completions, and hospitalizations, will be monitored as serious adverse events, and will be reported our hospital's IRB according to our Data Safety & Monitoring Plan. If a patient is deemed to need psychiatric hospitalization based on the screening, they will be withdrawn from the study.

That said, we will be clear during the assent/consent process with the parents and child that we will not be conducting ongoing, real-time monitoring of the text messaging. We will emphasize that if a child needs immediate assistance, s/he or his/her parents should call 911, the child's doctor, or call one of the crisis numbers provided.

By notifying parents/guardians of the teen's risk, providing parents with the information they need to monitor their child's risk, and by conducting ongoing monitoring of the safety of the teens, we are maintaining the highest ethical standard for our participants.

#### Risk 4) Violence

The emergence of increased aggression is important and needs to be monitored. If a subject discloses increasing frequency of involvement in violence, severe physical injury, homicidality, or high risk of retaliatory violence she will be contacted by the PI for further evaluation. Although no questions will be specifically asked about child abuse or sexual assault during the study, the staff will be trained to assess and respond to participants for whom these issues arise.

### **Risk 5) Mandatory Reporting and Crisis Management:**

As described above and in the Data Safety & Monitoring Plan, below, all instances of potential mental health or violence risks, staff will follow a written protocol regarding reporting these incidents to Dr. Ranney or Spirito based on call schedule, and will take appropriate referral or legal action as indicated. In addition, the IRB board at Rhode Island Hospital will be informed of any incidents. Drs. Ranney and Spirito will be responsible for providing training to all research staff who are conducting assessments with participants regarding procedures for identifying, managing, and responding appropriately to acute warning signs of distress that could occur as a result of the survey. Such strategies include maintaining an empathic response, acknowledging the distress through reflection, and eliciting or encouraging use of relaxation and cognitive

calming strategies. Staff will receive training in crisis assessment and management procedures in the event that participants reveal suicidal and/or homicidal ideation, child physical/sexual abuse, or concerns about safety. Drs. Ranney (M.D., Emergency Medicine) and Spirito (Ph.D., Clinical Psychology) will be responsible for providing regular supervision to research staff who have direct contact with patients including crisis procedures for suicide and homicide risk and clinical assessment and referral procedures for participants who are a danger to themselves or others. Supervision will focus on procedures for managing issues that could arise given the patient population, including potential crisis situations and/or adverse events.

Our crisis management procedures mirror those used by the Rhode Island Hospital Department of Psychiatry and Emergency Medicine clinical services. Dr. Ranney has successfully used these safety protocols in studies at the proposed study site.

It is possible that situations will arise in which researchers are provided with information by children or families which they are legally and ethically obligated to disclose (e.g., suicidal or homicidal intent, harsh disciplinary practices, sexual abuse). All participants are informed in advance through the process of informed consent of the legal and ethical obligations of study staff should these issues arise. The consent and assent forms will clearly describe times when confidentiality must be broken, i.e., suicidality, homicidal thoughts, and a report of child physical or sexual abuse. Participant confidentiality will be breached only to protect the safety and welfare of research participants and only in accordance with state and federal law.

As additional safeguards, if a child reveals substantial mental health problems, such as suicidal ideation/attempts, homicidal ideation, or clinical deterioration, or if such problems are identified during the course of the study, the child will be evaluated as soon as possible, by the PI, the primary mentor, and (if indicated) the on-call RIH psychiatric crisis team, to make a clinical determination about whether the child requires hospitalization or other clinical services. The primary mentor is a licensed child clinical psychologist and has training and experience in intervening in similar crisis situations. Project staff will carry cell phones with them during all participant contact and will be instructed to contact the PI (who is on call and always carries a phone) immediately to inform her of any clinical emergency. Additionally, Dr. Spirito and Dr. Ranney will carefully monitor the symptom progression of all participants. If a patient is deemed to need psychiatric hospitalization based on the screening, they will be withdrawn from the study.

If any mental health problems are reported or identified at the time of the follow-up and the family is not in treatment, appropriate referral for psychological intervention will be arranged.

Whenever possible, study staff will handle these situations therapeutically. For example, if time limits and safety concerns allow, parents will be informed in advance and provided the opportunity to participate in the mandated report process. Research staff will contact the PI who will be responsible for any on-site clinical decision-making.

Over the past 10 years, in several ED studies conducted by myself and my mentors, staff have encountered only 2 cases of harm to others that involved crisis management procedures leading to breaching confidentiality and involving authorities, less than 10 cases of child abuse requiring mandatory reporting to the police, and regular suicide risk assessments (~10 participants per study, per month).

### 14c. Potential benefits of the proposed research to the subjects and others:

Participation in this project could potentially benefit participants in a few important ways. The instruments used to obtain information in this study are commonly used in clinical and research practice but may invoke some emotional discomfort. Efforts will be made to minimize this discomfort by presenting questions in a supportive manner, assuring participants that they may refuse to answer questions that make them uncomfortable, and may terminate participation in the study at any time. It is also possible that the questions or assessments themselves may be beneficial to all participants by asking them to review their affect and peer violence. The screening and baseline assessments may therefore act as a very minimal intervention (as could any study with interviews regarding risky behaviors). Indeed, study participants in Dr. Spirito's and Dr. Cunningham's previous, similar studies have commented that they have found the questions to be helpful.

Additionally, we hope that our intervention will be successful in preventing/reducing depressive symptoms, and possibly peer violence, in our subject population. The intervention offers the possibility of a relatively low-resource, highly-disseminable preventive intervention for a needy population. We therefore think that the clear examination of these questions outweighs the previously mentioned risks.

Because all youth participating in the study self-report depressive symptoms and peer violence, we felt it was necessary to enhance usual care (typically no violence-prevention or mental health information is routinely provided during the ED visit) for all youth. Thus, all youth participating in screening will review a health information brochure, with referral information for mental health problems including suicide hotlines, substance

use, and violence prevention and treatment services, anger management, etc. This pamphlet will be similar in style and content to that used in my mentors' prior work. In addition, as described above, participants that meet criteria for severe depressive symptoms or suicidality on the screening survey will be offered a clinical assessment and individualized referral in the ED, which exceeds the current standard of care.

In sum, potential benefits for the research far outweigh the risks for the participants. The proposed research also has significant benefits for society in general, as described in **Importance of the Knowledge to be Gained** (14d, below).

## 14d. Importance of the Knowledge to be Gained

Given the high rates of both depression and peer violence among youth; the interdependence of these problems; the individual and societal cost of violence and its mental health consequences; the fact that most of these teens use the ED as their primary source of care; and these teens' lack of access to traditional mental health services; the development of effective targeted interventions are clearly needed. Given the paucity of accessible existing interventions, the knowledge to be gained from this research is significant. The risks to participants are reasonable in relation to the importance of this knowledge to be gained.

#### 14e. Vertebrate animals:

n/a

# 14f. Data and Safety Monitoring Plan

To address the NIH policy for Data and Safety Monitoring, the PI (Dr. Ranney) and her mentorship team have developed a system for oversight of the proposed study and its participants. The Data and Safety Monitoring Plan for this application will begin by implementing standard procedures for day-to-day monitoring of the study. The Principal Investigator, Dr. Ranney, will be responsible for monitoring the data quality and safety. As already noted above, all research projects involving human participants at Rhode Island Hospital, including this proposed study, require approvals from the Rhode Island Hospital (RIH)/Lifespan Institutional Review Board (IRB). In addition, because of the sensitive nature of the data being collected, a Certificate of Confidentiality will be obtained for this study from the National Institute of Health (NIH).

Dr. Ranney will ensure that all relevant IRB policies, procedures and stipulations are being followed. Dr Ranney also will be responsible for ensuring that other investigators and project staff adhere to the RIH IRB policies including the following: (1) All participants in the full Aim 2 and Aim 3 studies will understand, agree to, and sign a written assent form (and consent from parent/guardian) before participating; (2) Strict adherence to a participant's right to withdraw or refuse to answer questions will be maintained; (3) All interviews and assessments will be completely confidential and no names will be associated with the data; (4) Consent forms and identifying information will be kept separate from the actual participant data; (5) All identifying information (consents, tracking data) will be kept locked at all times and computer files will be saved with passwords; and (6) Participants will be informed in writing in the consent form on how to contact the PI, the study coordinator, and IRB office with any questions and/or concerns.

Weekly meetings with Dr. Spirito will be conducted to evaluate the progress of the trial and to review data quality, recruitment, study retention, and examine other factors that may affect outcome. Participant experiences and the rates of adverse events will also be reviewed to determine any changes in participant risk. Dr. Ranney will report any adverse events that are observed to the IRB within one week of occurrence, and to NIMH in our annual report. Serious adverse events (SAEs) will be reported to the IRB within 2 work days of our receipt of information regarding the event; if deemed to require a change in protocol, NIMH will also be notified. Reports of changes or amendments to the protocol in general must be requested first in writing to the IRB, which then will grant or deny permission to make the requested change or amendment in protocol.

Finally, if significant homicidal, suicidal, or mental health risks occur during the study period, the participant's parent(s) will be notified, as described in **14b.2**. **Protection against risks** (above), and evaluation by the Rhode Island Hospital crisis team will be immediately initiated to determine whether hospitalization is needed.

In the event that a research participant either withdraws from the study or the investigator decides to discontinue a research participant due to SAE, the research participant will be monitored by the investigator via ongoing status assessment until either a resolution is reached (i.e. the problem requiring hospitalization has resolved or stabilized with no further changes expected), the SAE is determined to be clearly unrelated to the study intervention, or the SAE results in death.

Independent evaluators from the Department of Emergency Medicine and the Department of Psychiatry will be incorporated into the existing Data Safety & Monitoring Board (DSMB) in the Department of Emergency

Medicine, to assist with study-specific ongoing monitoring of data. These additional members will include Dr. James Linakis (pediatric emergency physician and chair of the Lifespan IRB, Dept of EM, Brown University); and Dr. Michael J. Mello (emergency physician and researcher in the overlap between alcohol abuse and injury, Dept of EM, Brown University). This enhanced Dept of EM DSMB, as an adjunct to the IRB, will have control and independence in offering recommendation arising from participant concerns or adverse events related to our study, or stopping the study for the benefit of our participants. This DSMB will convene once yearly, and as needed, and produce a written report. This report will be sent to the Lifespan IRB as well as to the project officer at NIMH. The DSMB will review all serious or unexpected adverse events to determine any changes in participant risk and provide recommendations.

Participants will only be identified by number during review of study progress by the DSMB. In the event that confidentiality must be breached, only the PI and Primary Mentors would be informed of identifying information in order to report to the appropriate authorities or health care providers. In the event that a conflict of interest within the DSMB is identified, the DSMB will disclose the matter to the Lifespan IRB. The DSMB will provide recommendations to the PI on how to resolve the conflict of interest, and the PI will report and document the action to the Lifespan IRB.

## 14g. Educational Training

Since October 1, 2001, Lifespan has required that researchers and IRB members read Protecting Study Volunteers in Research (Dunn & Chadwick) and complete the related exam. This process has served as initial certification between 10/2001 and 5/2005. In June, 2005, the Office of Research Administration contracted with CITI, a Collaborative Institutional (modular) Training Initiative program, for our Human Subjects protection and HIPAA training for all research personnel. Currently this program offers our researchers a basic human subject's protection course as well as a refresher course which we require every three years. Documentation of successful completion is automatically generated and should be printed directly by the researcher. For further information regarding Lifespan's Human Subject's Protection course go to: http://www.lifespan.org/research/IRB/MandatoryEdguidance.asp

Additional and continuing education opportunities for clinical researchers include the Office of Research Administration newsletter that is circulated to > 900 recipients every 6 weeks. Relevant information concerning research review is available on the ORA web page at www2.lifespan.org/research/. In addition to standard institutional research information, the web page contains links to other sites such as CenterWatch, NIH, PRIM&R/ARENA.

Finally, the PI will participate in the training in the Responsible Conduct of Research detailed in Section 5, above.

- 1. Hawker DSJ, Boulton MJ. Twenty years' research on peer victimization and psychosocial maladjustment: a meta-analytic review of cross-sectional studies. J Child Psychol Psychiatry 2000;41(4):441-455.
- 2. Obeidallah DA, Earls FJ. Adolescent Girls: The Role of Depression in the Development of Delinquency. Washington, DC: National Institute of Justice, 1999.
- 3. Ford JD, Elhai JD, Connor DF, et al. Poly-victimization and risk of posttraumatic, depressive, and substance use disorders and involvement in delinquency in a national sample of adolescents. J Adolesc Health 2010;46(6):545-552.
- 4. Pailler ME, Kassam-Adams N, Datner EM, et al. Depression, acute stress and behavioral risk factors in violently injured adolescents. Gen Hosp Psychiatry 2007 Jul-Aug;29(4):357-363.
- 5. Saluja G, Iachan R, Scheidt PC, et al. Prevalence of and risk factors for depressive symptoms among young adolescents. Arch Pediatr Adolesc Med 2004 Aug;158(8):760-765.
- 6. Wade TJ, Cairney JP, Pevalin DJ. Emergence of gender differences in depression during adolescence: National panel results from three countries. J Am Acad Child Adolesc Psychiatry 2002;41(2):190-198.
- 7. Lewinsohn PM, Hops H, Roberts RE, et al. Adolescent psychopathology: I. Prevalence and incidence of depression and other DSM-III-R disorders in high school students. J Abnorm Psychol 1993 Feb;102(1):133-144.
- 8. Rutman MS, Shenassa E, Becker BM. Brief screening for adolescent depressive symptoms in the emergency department. Acad Emerg Med 2008 Jan;15(1):17-22.

- 9. Ranney ML, Whiteside L, Walton MA, et al. Sex differences in characteristics of adolescents presenting to the emergency department with acute assault-related injury. Acad Emerg Med 2011 Oct;18(10):1027-1035.
- 10. Seiffge-Krenke I. Causal links between stressful events, coping style, and adolescent symptomatology. J Adolesc 2000 Dec;23(6):675-691.
- 11. Bell CC, McBride DF. Affect regulation and prevention of risky behaviors. JAMA 2010 August 4, 2010;304(5):565-566.
- 12. Hankin BL, Abramson LY. Development of gender differences in depression: An elaborated cognitive vulnerability-transactional stress theory. Psychol Bull 2001 Nov;127(6):773-796.
- 13. Herts KL, McLaughlin KA, Hatzenbuehler ML. Emotion dysregulation as a mechanism linking stress exposure to adolescent aggressive behavior. J Abnorm Child Psychol 2012 Mar 31.
- 14. Cuevas CA, Finkelhor D, Clifford C, et al. Psychological distress as a risk factor for revictimization in children. Child Abuse Negl 2010 Mar 19.
- 15. Cuevas CA, Finkelhor D, Ormrod R, et al. Psychiatric diagnosis as a risk marker for victimization in a national sample of children. J Interpers Violence 2009 Apr;24(4):636-652.
- 16. Fergusson DM, Lynskey MT, Horwood LJ. Origins of comorbidity between conduct and affective disorders. J Am Acad Child Adolesc Psychiatry 1996;35(4):451-460.
- 17. Ferguson CJ, San Miguel C, Hartley RD. A multivariate analysis of youth violence and aggression: The influence of family, peers, depression, and media violence. J Pediatr 2009 Dec;155(6):904-908 e903.
- 18. Robinson WL, Paxton KC, Jonen LP. Pathways to aggression and violence among African American adolescent males: the influence of normative beliefs, neighborhood, and depressive symptomatology. J Prev Interv Community 2011 Apr;39(2):132-148.
- 19. McLaughlin KA, Hatzenbuehler ML, Hilt LM. Emotion dysregulation as a mechanism linking peer victimization to internalizing symptoms in adolescents. J Consult Clin Psychol 2009 Oct;77(5):894-904.
- 20. Dempsey M. Negative coping as mediator in the relation between violence and outcomes: Inner-city African American youth. Am J Orthopsychiatry 2002 Jan;72(1):102-109.
- 21. Berkowitz SJ. Children exposed to community violence: The rationale for early intervention. Clin Child Fam Psychol Rev 2003 Dec;6(4):293-302.
- 22. Lambert SF, Copeland-Linder N, Ialongo NS. Longitudinal associations between community violence exposure and suicidality. J Adolesc Health 2008 Oct;43(4):380-386.
- 23. O'Donnell L, Stueve A, Wilson-Simmons R. Aggressive behaviors in early adolescence and subsequent suicidality among urban youths. J Adolesc Health 2005 Dec;37(6):517.
- 24. Luk JW, Wang J, Simons-Morton BG. Bullying victimization and substance use among U.S. adolescents: Mediation by depression. Prev Sci 2010 Dec;11(4):355-359.
- 25. D'Onofrio G, Jauch E, Jagoda A, et al. NIH roundtable on opportunities to advance research on neurologic and psychiatric emergencies. Ann Emerg Med 2010 Nov;56(5):551-564.
- 26. Rhodes KV, Gordon JA, Lowe RA. Preventive care in the emergency department, part I: Clinical preventive services; are they relevant to Emergency Medicine? Acad Emerg Med 2000;7(9):1036-1041.
- 27. Cunningham R, Knox L, Fein J, et al. Before and after the trauma bay: The prevention of violent injury among youth. Ann Emerg Med 2009;53(4):490-500.
- 28. Stein BD, Jaycox LH, Kataoka SH, et al. A mental health intervention for schoolchildren exposed to violence: a randomized controlled trial. JAMA 2003 August 6, 2003;290(5):603-611.
- 29. Kataoka SH, Stein BD, Jaycox LH, et al. A school-based mental health program for traumatized Latino immigrant children. J Am Acad Child Adolesc Psychiatry 2003 Mar;42(3):311-318.
- 30. Merikangas KR, He JP, Burstein M, et al. Service utilization for lifetime mental disorders in U.S. adolescents: results of the National Comorbidity Survey-Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry 2011 Jan;50(1):32-45.
- 31. Wilson KM, Klein JD. Adolescents who use the emergency department as their usual source of care. Arch Pediatr Adolesc Med 2000 April 1, 2000;154(4):361-365.

- 32. Sabin JA, Zatzick DF, Jurkovich G, et al. Primary care utilization and detection of emotional distress after adolescent traumatic injury: Identifying an unmet need. Pediatrics 2006 January 1, 2006;117(1):130-138.
- 33. Cummings JR, Druss BG. Racial/ethnic differences in mental health service use among adolescents with major depression. J Am Acad Child Adolesc Psychiatry 2011;50(2):160-170.
- 34. Cohen JA. Early mental health interventions for trauma and traumatic loss in children and adolescents. In: Litz BT, ed. Early Interventions for Trauma and Traumatic Loss. New York, NY: Guilford Press, 2004:131-146.
- 35. Rhodes KV. Mood disorders in the emergency department: The challenge of linking patients to appropriate services. Gen Hosp Psychiatry 2008 Jan-Feb;30(1):1-3.
- 36. Baren JM, Mace SE, Hendry PL, et al. Children's mental health emergencies-part 1: Challenges in care: Definition of the problem, barriers to care, screening, advocacy, and resources. Pediatr Emerg Care 2008 Jun;24(6):399-408.
- 37. Lenhart A, Ling R, Campbell S, et al. Teens and mobile phones. Pew Internet and American Life Project 2010 [cited April 20, 2010]; Available from: http://pewinternet.org/~/media//Files/Reports/2010/PIP-Teens-and-Mobile-2010.pdf
- 38. Fjeldsoe BS, Marshall AL, Miller YD. Behavior change interventions delivered by mobile telephone short-message service. Am J Prev Med 2009 Feb;36(2):165-173.
- 39. Whittaker R, Merry S, Stasiak K, et al. MEMO A mobile phone depression prevention intervention for adolescents: development process and postprogram findings on acceptability from a randomized controlled trial. J Med Internet Res 2012;14(1):e13.
- 40. Heron KE, Smyth JM. Ecological momentary interventions: Incorporating mobile technology into psychosocial and health behaviour treatments. Br J Health Psychol 2010 Feb;15(Pt 1):1-39.
- 41. National Institutes of Health. NIH Science of Behavior Change, June 15-16, 2009.; 2009; Bethesda, MD; 2009.
- 42. Cunningham RM, Chermack ST, Zimmerman MA, et al. Brief motivational interviewing intervention for peer violence and alcohol use in teens: one-year follow-up. Pediatrics 2012 May 21.
- 43. Stice E, Rohde P, Gau JM, et al. Efficacy trial of a brief cognitive-behavioral depression prevention program for high-risk adolescents: Effects at 1- and 2-year follow-up. J Consult Clin Psychol 2010 Sep 27;78(6):856-867.
- 44. Walton M, Chermack S, Shope J, et al. Effects of a brief intervention for reducing violence and alcohol misuse among adolescents: A randomized trial. JAMA 2010 2010;304(5):527-535.
- 45. Zatzick D, Jurkovich G, Rivara F, et al. A randomized stepped care intervention trial targeting posttraumatic stress disorder for surgically hospitalized injury survivors. Ann Surg 2012;IN PRESS.
- 46. National Institute of Mental Health. From Discovery to Cure: Acceleration the Development of New and Personalized Interventions for Mental Illness; August 2010.
- 47. Spirito A, Monti PM, Barnett NP, et al. A randomized clinical trial of a brief motivational intervention for alcohol-positive adolescents treated in an emergency department. J Pediatr 2004;145(3):396-402.
- 48. Attkisson CC, Zwick R. The Client Satisfaction Questionnaire: Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann 1982;5(3):233-237.
- 49. Young JE, Beck AT. Cognitive Therapy Scale Rating Manual. Philadelphia, PA: Center for Cognitive Therapy, 1980.
- 50. Moyers TB, Martin T, Manuel JK, et al. Assessing competence in the use of motivational interviewing. J Subst Abuse Treat 2005;28(1):19-26.
- 51. Resko SM, Walton MA, Chermack ST, et al. Therapist competence and treatment adherence for a brief intervention addressing alcohol and violence among adolescents. J Subst Abuse Treat 2012 Jun;42(4):429-437.
- 52. Hollon SD, Muñoz RF, Barlow DH, et al. Psychosocial intervention development for the prevention and treatment of depression: Promoting innovation and increasing access. Biol Psych 2002;52(6):610-630.

- 53. NIH State-of-the-Science Conference Statement on preventing violence and related health-risking social behaviors in adolescents. NIH Consens State Sci Statements 2004 Oct 13-15;21(2):1-34.
- 54. Preventing mental, emotional, and behavioral disorders among young people: progress and possibilities. Committee on Prevention of Mental Disorders and Substance Abuse Among Children, Youth, and Young Adults: Research Advances and Promising Interventions. Washington, DC: National Academies Press, 2009.
- 55. U.S. Department of Health and Human Services. Healthy People 2020: Topics and Objectives. 2010 [cited July 9, 2012]; Available from:

http://www.healthypeople.gov/2020/topicsobjectives2020/default.aspx

- 56. Merikangas KR, He J, Burstein M, et al. Lifetime prevalence of mental disorders in U.S. adolescents: Results from the National Comorbidity Survey Replication-Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry 2010;49(10):980-989.
- 57. Goldstein AL, Walton MA, Cunningham RM, et al. Violence and substance use as risk factors for depressive symptoms among adolescents in an urban emergency department. J Adolesc Health 2007 Mar;40(3):276-279.
- 58. Graves KN. Not always sugar and spice: Expanding theoretical and functional explanations for why females aggress. Aggress Violent Behav 2007;12(2):131-140.
- 59. Zatzick DF, Jurkovich GJ, Fan M-Y, et al. Association between posttraumatic stress and depressive symptoms and functional outcomes in adolescents followed up longitudinally after injury hospitalization. Arch Pediatr Adolesc Med 2008 July 1, 2008;162(7):642-648.
- 60. Eaton DK, Kann L, Kinchen S, et al. Youth risk behavior surveillance United States, 2011. MMWR Surveill Summ 2012 Jun 8;61(4):1-162.
- 61. Youth violence: Facts at a glance. 2010 [cited 2012 July 9]; Available from: <a href="http://www.cdc.gov/violenceprevention/pdf/YV-DataSheet-a.pdf">http://www.cdc.gov/violenceprevention/pdf/YV-DataSheet-a.pdf</a>
- 62. CDC. Web-based Injury Statistics Query and Reporting System (WISQARS™). US Department of Health and Human Services, Centers for Disease Control and Prevention.
- 63. Biros MH, Hick K, Cen YY, et al. Occult depressive symptoms in adolescent emergency department patients. Arch Pediatr Adolesc Med 2008 Aug;162(8):769-773.
- 64. Ranney ML, Choo EK, Spirito A, et al. Adolescents' preference for technology-based emergency department behavioral interventions, according to self-reported risky behaviors. Pediatr Emerg Care 2012;UNDER REVIEW.
- 65. Ranney ML, Walton M, Zimmerman M, et al. Depressive symptoms among youth with a history of peer violence: a gender-stratified analysis. Gen Hosp Psychiatry 2012;UNDER REVIEW.
- 66. Kessler RC, Walters EE. Epidemiology of DSM-III-R major depression and minor depression among adolescents and young adults in the national comorbidity survey. Depress Anxiety 1998;7(1):3-14.
- 67. Nicolaidis C, Curry M, McFarland B, et al. Violence, mental health, and physical symptoms in an academic internal medicine practice. J Gen Intern Med 2004 Aug;19(8):819-827.
- 68. Margolin G, Vickerman KA, Oliver PH, et al. Violence exposure in multiple interpersonal domains: Cumulative and differential effects. J Adolesc Health 2010 Aug;47(2):198-205.
- 69. Seeley JR, Stice E, Rohde P. Screening for depression prevention: Identifying adolescent girls at high risk for future depression. J Abnorm Psychol 2009 Feb;118(1):161-170.
- 70. Nicolaidis C. Violence and poor mental health and functional outcomes. Bmj 2011;343:d7311.
- 71. Bernstein SL. The clinical impact of health behaviors on emergency department visits. Acad Emerg Med 2009;16(11):1054-1059.
- 72. Bernstein SL, D'Onofrio G. Public health in the emergency department: *Academic Emergency Medicine* consensus conference executive summary. Acad Emerg Med 2009;16(11):1037-1039.
- 73. Cyranowski JM, Frank E, Young E, et al. Adolescent onset of the gender difference in lifetime rates of major depression: A theoretical model. Arch Gen Psychiatry 2000 January 1, 2000;57(1):21-27.

- 74. Borowsky IW, Ireland M. Predictors of future fight-related injury among adolescents. Pediatrics 2004 Mar;113(3 Pt 1):530-536.
- 75. Marcus RF. Cross-sectional study of violence in emerging adulthood. Aggress Behav 2009 03;35(2):188-202.
- 76. Copeland-Linder N, Lambert SF, Ialongo NS. Community violence, protective factors, and adolescent mental health: A profile analysis. J Clin Child Adolesc Psychol 2010;39(2):176 186.
- 77. Lipschitz DS, Rasmusson AM, Anyan W, et al. Clinical and functional correlates of posttraumatic stress disorder in urban adolescent girls at a primary care clinic. J Am Acad Child Adolesc Psychiatry 2000 Sep;39(9):1104-1111.
- 78. Carter JS, Grant KE. A prospective comparison of moderating relationships among stressors, hopelessness, and internalizing symptoms in low-income urban youth with asthma. J Urban Health 2012 Jun 7.
- 79. Kort-Butler LA. Coping styles and sex differences in depressive symptoms and delinquent behavior. J Youth Adolesc 2009 Jan;38(1):122-136.
- 80. Kelly EG, Kelly LG, Jeremy WP, et al. Problem solving moderates the effects of life event stress and chronic stress on suicidal behaviors in adolescence. J Clin Psychol 2009;65(12):1281-1290.
- 81. Merry S, McDowell H, Wild CJ, et al. A randomized placebo-controlled trial of a school-based depression prevention program. J Am Acad Child Adolesc Psychiatry 2004 May;43(5):538-547.
- 82. Stice E, Rohde P, Seeley JR, et al. Brief cognitive-behavioral depression prevention program for high-risk adolescents outperforms two alternative interventions: A randomized efficacy trial. J Consult Clin Psychol 2008 Aug;76(4):595-606.
- 83. Garber J, Clarke GN, Weersing VR, et al. Prevention of depression in at-risk adolescents: A randomized controlled trial. JAMA 2009 Jun 3;301(21):2215-2224.
- 84. Stice E, Shaw H, Bohon C, et al. A meta-analytic review of depression prevention programs for children and adolescents: Factors that predict magnitude of intervention effects. J Consult Clin Psychol 2009 Jun;77(3):486-503.
- 85. Clarke GN, Hawkins W, Murphy M, et al. Targeted prevention of unipolar depressive disorder in an at-risk sample of high school adolescents: a randomized trial of a group cognitive intervention. J Am Acad Child Adolesc Psychiatry 1995 Mar;34(3):312-321.
- 86. Cunningham RM, Walton MA, Goldstein AL, et al. Three-month follow-up of brief computerized and therapist interventions for alcohol and violence among teens. Acad Emerg Med 2009;16(11):1193-1207.
- 87. Snider CE, Lee JS. Emergency department dispositions among 4100 youth injured by violence: A population-based study. CJEM 2007 May;9(3):164-169.
- 88. Bisgaier J, Rhodes KV. Auditing access to specialty care for children with public insurance. N Engl J Med 2011 Jun 16;364(24):2324-2333.
- 89. Spirito A, Boergers J, Donaldson D, et al. An intervention trial to improve adherence to community treatment by adolescents after a suicide attempt. J Am Acad Child Adolesc Psychiatry 2002 Apr;41(4):435-442.
- 90. Pailler ME, Cronholm PF, Barg FK, et al. Patients' and caregivers' beliefs about depression screening and referral in the emergency department. Pediatr Emerg Care 2009 November;25(11):721-727.
- 91. Horowitz JL, Garber J. The prevention of depressive symptoms in children and adolescents: A meta-analytic review. J Consult Clin Psychol 2006 Jun;74(3):401-415.
- 92. Fleischmann A, Bertolote JM, Wasserman D, et al. Effectiveness of brief intervention and contact for suicide attempters: a randomized controlled trial in five countries. Bulletin of the World Health Organization 2008;86:703-709.
- 93. Carter GL, Clover K, Whyte IM, et al. Postcards from the EDge: 24-month outcomes of a randomised controlled trial for hospital-treated self-poisoning. Br J Psychiatry 2007 Dec;191:548-553.

- 94. Vaiva G, Vaiva G, Ducrocq F, et al. Effect of telephone contact on further suicide attempts in patients discharged from an emergency department: randomised controlled study. BMJ 2006 May 27;332(7552):1241-1245.
- 95. Ranney ML, Choo EK, Wang Y, et al. Emergency department patients' preferences for technology-based behavioral interventions. Ann Emerg Med 2012 Apr 26;IN PRESS.
- 96. Depp CA, Mausbach B, Granholm E, et al. Mobile interventions for severe mental illness: design and preliminary data from three approaches. J Nerv Ment Dis 2010 Oct;198(10):715-721.
- 97. Morris ME, Kathawala Q, Leen TK, et al. Mobile therapy: Case study evaluations of a cell phone application for emotional self-awareness. J Med Internet Res 2010;12(2):e10.
- 98. Hyden C, Cohall A. Innovative approaches to using new media and technology in health promotion for adolescents and young adults. Adolesc Med State Art Rev 2011 Dec;22(3):498-520, xi-xii.
- 99. Rizvi SL, Dimeff LA, Skutch J, et al. A pilot study of the DBT coach: an interactive mobile phone application for individuals with borderline personality disorder and substance use disorder. Behav Ther 2011 Dec;42(4):589-600.
- 100. Ahmead M, Bower P. The effectiveness of self help technologies for emotional problems in adolescents: A systematic review. Child Adolesc Psychiatry Ment Health 2008;2(1):20.
- 101. Agyapong VI, Ahern S, McLoughlin DM, et al. Supportive text messaging for depression and comorbid alcohol use disorder: single-blind randomised trial. J Affect Disord 2012 Mar 28.
- 102. Free C, Knight R, Robertson S, et al. Smoking cessation support delivered via mobile phone text messaging (txt2stop): A single-blind, randomised trial. Lancet 2011 Jul 2;378(9785):49-55.
- 103. Granholm E, Ben-Zeev D, Link PC, et al. Mobile Assessment and Treatment for Schizophrenia (MATS): a pilot trial of an interactive text-messaging intervention for medication adherence, socialization, and auditory hallucinations. Schizophr Bull 2011 Nov 10.
- 104. Suffoletto B, Callaway C, Kristan J, et al. Text-message-based drinking assessments and brief interventions for young adults discharged from the emergency department. Alcohol Clin Exp Res 2012 Mar;36(3):552-560.
- 105. Arora S, Peters AL, Agy C, et al. A mobile health intervention for inner city patients with poorly controlled diabetes: Proof-of-concept of the TExT-MED program. Diabetes Technol Ther 2012 Apr 23.
- 106. Boyer EW, Fletcher R, Fay RJ, et al. Preliminary efforts directed toward the detection of craving of illicit substances: The iHeal Project. J Med Toxicol 2012 Feb 4.
- 107. Boyer EW, Picard RW. A mobile enabling technology to promote adherence to behavioral therapy. University of Massachusetts Medical School, Worcester, MA: National Institute on Drug Abuse, RC1DA028428-01 2009-2011.
- 108. Cunningham RM. Substance Use among Violently Injured Youth in an Urban ER: Services and Outcomes. University of Michigan, Ann Arbor, MI: National Institute on Drug Abuse, R01DA024646-02 2009.
- 109. Walton MA, Cunningham RM. Optimizing Brief Alcohol Intervention for Underage Drinkers in the ER. University of Michigan, Ann Arbor, MI: National Institue on Alcohol Abuse and Alcoholism, 2009.
- 110. Linakis JG, Spirito A. ED Based Prevention Intervention to Delay Alcohol Use by Young Adolescents. Rhode Island Hospital/Alpert Medical School, Brown University, Providence, RI: National Institue on Alcohol Abuse and Alcoholism, R21AA018380-01A1 2010.
- 111. Whittaker R, Maddison R, McRobbie H, et al. A multimedia mobile phone-based youth smoking cessation intervention: Findings from content development and piloting studies. J Med Internet Res 2008;10(5):e49.
- 112. Spirito A, Sindelar-Manning H, Colby SM, et al. Individual and family motivational interventions for alcohol-positive adolescents treated in an emergency department: results of a randomized clinical trial. Arch Pediatr Adolesc Med 2011 Mar;165(3):269-274.

- 113. Bearman PS, Jones J, Udry JR. The National Longitudinal Study of Adolescent Health: Research Design [online]. . 1997 [cited; Available from:
- http://www.cpc.unc.edu/projects/addhealth/design.html
- 114. Cunningham R, Walton M, Trowbridge M, et al. Correlates of violent behavior among adolescents presenting to an urban emergency department. J Pediatr 2006 Dec;149(6):770-776.
- 115. Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Appl Psychol Meas 1977 June 1, 1977;1(3):385-401.
- 116. Straus MA, Hamby SL, Boney-McCoy S, et al. The revised conflict tactics scales (CTS2): Development and preliminary psychometric data. J Fam Issues 1996;17(3):283-316.
- 117. Radloff LS. The use of the Center for Epidemiologic Studies Depression Scale in adolescents and young adults. J Youth Adolesc 1991;20(2):149-166.
- 118. Asarnow JR, Jaycox LH, Duan N, et al. Effectiveness of a quality improvement intervention for adolescent depression in primary care clinics: A randomized controlled trial. JAMA 2005 Jan 19;293(3):311-319.
- 119. Wilcox H, Field T, Prodromidis M, et al. Correlations between the BDI and CES-D in a sample of adolescent mothers. Adolescence 1998 Fall;33(131):565-574.
- 120. Garrison CZ, Addy CL, Jackson KL, et al. The CES-D as a screen for depression and other psychiatric disorders in adolescents. J Am Acad Child Adolesc Psychiatry 1991 Jul;30(4):636-641.
- 121. Dierker LC, Albano AM, Clarke GN, et al. Screening for anxiety and depression in early adolescence. J Am Acad Child Adolesc Psychiatry 2001 Aug;40(8):929-936.
- 122. Whiteside L, Ranney ML, Chermack ST, et al. The overlap of youth violence among aggressive adolescents with past year alcohol use, a latent class analysis: aggression and victimization in peer and dating violence in an inner city emergency department. J Stud Alcohol Drugs 2012;UNDER REVISION.
- 123. Usability Guidelines. [cited July 9, 2012]; Available from: http://usability.gov/guidelines/index.html
- 124. Brooke J. System Usability Scale. 1986 [cited June 5, 2012]; Available from: <a href="http://usability.gov/templates/index.html">http://usability.gov/templates/index.html</a>
- 125. Bangor A, Kortum PT, Miller JT. An empirical evaluation of the System Usability Scale. Int J Human-Computer Interaction 2008 2008/07/29;24(6):574-594.
- 126. Lewis JR, Sauro J. The factor structure of the System Usability Scale. Proceedings of the 1st International Conference on Human Centered Design: Held as Part of HCI International 2009. San Diego, CA: Springer-Verlag, 2009:94-103.
- 127. Picard RW, Liu KK. Relative subjective count and assessment of interruptive technologies applied to mobile monitoring of stress. International Journal of Human-Computer Studies 2007;65(4):361-375.
- 128. Liu KK. A Personal, Mobile System for Understanding Stress and Interruptions. Boston, MA: MIT Media Arts and Science; 2004.
- 129. Rounsaville B, Carroll KM. A stage model of behavioral therapies research: Getting started and moving on from Stage I. Clin Psychol 2001;8(2):133-142.
- 130. Beck AT, Steer RA, Carbin MG. Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clinical Psychology Review 1988;8(1):77-100.
- 131. Bennett DS, Ambrosini PJ, Bianchi M, et al. Relationship of Beck Depression Inventory factors to depression among adolescents. J Affect Disord 1997 Sep;45(3):127-134.
- 132. Wolfe DA, Scott K, Reitzel-Jaffe D, et al. Development and validation of the Conflict in Adolescent Dating Relationships Inventory. Psychol Assess 2001 06;13(2):277-293.
- 133. Beck AT, Steer RA. Beck Anxiety Inventory Manual. San Antonio, TX: Psychological Corporation, 1993.
- 134. Foa EB, Johnson KM, Feeny NC, et al. The Child PTSD Symptom Scale: A preliminary examination of its psychometric properties. J Clin Child Psychol 2001 Sep;30(3):376-384.
- 135. Ascher BH, Farmer EMZ, Burns BJ, et al. The Child and Adolescent Services Assessment (CASA): Description and psychometrics. J Emot Behav Disord 1996;4(1):12-20.

- 136. Calvete E, Cardenoso O. Gender differences in cognitive vulnerability to depression and behavior problems in adolescents. J Abnorm Child Psychol 2005 Apr;33(2):179-192.
- 137. Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann 1982;5(3):233-237.
- 138. Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res 2011 May;45(5):626-629.
- 139. Kraemer HC, Mintz J, Noda A, et al. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry 2006 May;63(5):484-489.
- 140. Graham JW. Missing data analysis: Making it work in the real world. Annu Rev Psychol 2009;60:549-576.
- 141. Chambless DL, Hollon SD. Defining empirically supported therapies. J Consult Clin Psychol 1998 Feb;66(1):7-18.
- 142. Rogosa D, Brandt D, Zimowski M. A growth curve approach to the measurement of change. Psychol Bull 1982;92(3):726-748.
- 143. Zeger SL, Liang KY, Albert PS. Models for longitudinal data: A generalized estimating equation approach. Biometrics 1988 Dec;44(4):1049-1060.
- 144. Little RJ, Rubin DB. Statistical Analysis with Missing Data, 2nd edition. Hoboken, NJ: Wiley Interscience, 2002.
- 145. Graham J, Schafer J. Statistical strategies for small sample research. Thousand Oaks, CA: Sage, 1999.
- 146. Aarons GA, Covert J, Skriner LC, et al. The eye of the beholder: youths and parents differ on what matters in mental health services. Adm Policy Ment Health 2010 Nov;37(6):459-467.
- 147. Harris Interactive. A Generation Unplugged Research Report. 2008 [cited July 9, 2012]; Available from: <a href="http://files.ctia.org/pdf/HI">http://files.ctia.org/pdf/HI</a> TeenMobileStudy ResearchReport.pdf
- 148. Zickhur K. Generations and Their Gadgets. Washington DC: Pew Research Center; 2011.
- 149. Ranney ML, Verhoek-Oftedahl W, Rommel J, et al. Analysis of intentional and unintentional injuries caused by firearms and cutting/piercing instruments among Providence youth, Nov 2004-Dec 2007. Med Health R I 2009 Jun;92(6):200-203.
- 150. Ranney ML, Mello MJ. 433: Chart Review of Female Versus Male Adolescent Victims of Violence Presenting to the Emergency Department, 2004-2007. Ann Emerg Med 2010;56(3):S140.
- 151. Santelli JS, Smith Rogers A, Rosenfeld WD, et al. Guidelines for adolescent health research: A position paper of the Society for Adolescent Medicine. J Adolesc Health 2003;33(5):396-409.
- 152. Broderick J, Vikingstad G. Frequent assessment of negative symptoms does not induce depressed mood. J Clin Psychol Med Settings 2008;15(4):296-300.
- 153. Granholm E, Loh C, Swendsen J. Feasibility and validity of computerized ecological momentary assessment in schizophrenia. Schizophr Bull 2008 May 1, 2008;34(3):507-514.
- 154. Gwaltney CJ, Bartolomei R, Colby SM, et al. Ecological momentary assessment of adolescent smoking cessation: A feasibility study. Nicotine Tob Res 2008 Jul;10(7):1185-1190.
- 155. Weitzel JA, Bernhardt JM, Usdan S, et al. Using wireless handheld computers and tailored text messaging to reduce negative consequences of drinking alcohol. J Stud Alcohol Drugs 2007 Jul;68(4):534-537.
- 156. Bjorling EA. The momentary relationship between stress and headaches in adolescent girls. Headache 2009 Sep;49(8):1186-1197.
- 157. Delespaul PA, deVries MW. The daily life of ambulatory chronic mental patients. J Nerv Ment Dis 1987 Sep;175(9):537-544.
- 158. Epstein DH, Willner-Reid J, Vahabzadeh M, et al. Real-time electronic diary reports of cue exposure and mood in the hours before cocaine and heroin craving and use. Arch Gen Psychiatry 2009 Jan:66(1):88-94.
- 159. Freedman MJ, Lester KM, McNamara C, et al. Cell phones for ecological momentary assessment with cocaine-addicted homeless patients in treatment. J Subst Abuse Treat 2006 Mar;30(2):105-111.

- 160. Helgeson VS, Lopez LC, Kamarck T. Peer relationships and diabetes: Retrospective and ecological momentary assessment approaches. Health Psychol 2009 May;28(3):273-282.
- 161. Lukasiewicz M, Fareng M, Benyamina A, et al. Ecological momentary assessment in addiction. Expert Rev Neurother 2007 Aug;7(8):939-950.
- 162. Nock MK, Prinstein MJ, Sterba SK. Revealing the form and function of self-injurious thoughts and behaviors: A real-time ecological assessment study among adolescents and young adults. J Abnorm Psychol 2009 Nov;118(4):816-827.
- 163. Tasca GA, Illing V, Balfour L, et al. Psychometric properties of self-monitoring of eating disorder urges among treatment seeking women: Ecological momentary assessment using a daily diary method. Eat Behav 2009 Jan;10(1):59-61.
- 164. Head KJ, Noar SM, Iannarino NT, et al. Efficacy of text messaging-based interventions for health promotion: A meta-analysis. Social Science & Medicine 2013;97(0):41-48.
- 165. Kauer SD, Reid SC, Crooke AH, et al. Self-monitoring using mobile phones in the early stages of adolescent depression: randomized controlled trial. J Med Internet Res 2012;14(3):e67.
- 166. Suffoletto B, Akers A, McGinnis KA, et al. A Sex Risk Reduction Text-Message Program for Young Adult Females Discharged From the Emergency Department. J Adolesc Health 2013 May 23;53(3):387-393.
- 167. Hingle M, Nichter M, Medeiros M, et al. Texting for health: the use of participatory methods to develop healthy lifestyle messages for teens. J Nutr Educ Behav 2013 Jan-Feb;45(1):12-19.
- 168. Militello LK, Kelly SA, Melnyk BM. Systematic review of text-messaging interventions to promote healthy behaviors in pediatric and adolescent populations: implications for clinical practice and research. Worldviews Evid Based Nurs 2012 Apr;9(2):66-77.
- 169. Karasz HN, Eiden A, Bogan S. Text Messaging to Communicate With Public Health Audiences: How the HIPAA Security Rule Affects Practice. Am J Public Health 2013 Feb 14;IN PRESS.